CLINICAL TRIAL: NCT03664531
Title: Crossover Trial of Gluten and Gluten With Amylase-trypsin Inhibitors as Triggers of Gastrointestinal Symptoms in Patients With Irritable Bowel Syndrome
Brief Title: Dietary Triggers of Gastrointestinal Symptoms in IBS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Premysl Bercik, MD, Associate Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Diet in IBS
Record Dates: First submitted 2018-08-22; First posted 2018-09-10 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: crossover; gluten; amylase trypsin inhibitors; diet; challenge
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Nocebo Effect

STUDY DESIGN:
Intervention Model Description: Participants will be required to be on a gluten-free diet for a period of 3 weeks before starting the study. Participants will then be randomized to take muesli bars containing either purified gluten, non-purified gluten with amylase trypsin inhibitors, or nocebo for 1 week followed by 2 weeks of washout, and then repeated for the two remaining dietary challenges so that at the end all participants have been on all dietary challenges. At the beginning and end of each challenge period, participants will visit the clinic to be evaluated for changes in IBS symptoms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The statistician will also be masked from the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Gluten, ATIs, nocebo (Experimental): Participants will start on 1 week of muesli bars with purified gluten followed by 14 days washout. They will then take 1 week of muesli bars with non-purified gluten (containing ATIs) followed by 14 days of washout. Finally, they will have 1 week of nocebo muesli bars (with nothing).
  Interventions: Other: Purified gluten; Other: Non-purified gluten (containing ATIs); Other: Nocebo
- Gluten, nocebo, ATIs (Experimental): Participants will start on 1 week of muesli bars with purified gluten followed by 14 days washout. They will then take 1 week of nocebo muesli bars (with nothing) followed by 14 days of washout. Finally, they will have 1 week of muesli bars with non-purified gluten (containing ATIs).
  Interventions: Other: Purified gluten; Other: Non-purified gluten (containing ATIs); Other: Nocebo
- ATIs, gluten, nocebo (Experimental): Participants will start on 1 week of muesli bars with non-purified gluten (containing ATIs) followed by 14 days washout. They will then take 1 week of muesli bars with purified gluten followed by 14 days of washout. Finally, they will have 1 week of nocebo muesli bars (with nothing).
  Interventions: Other: Purified gluten; Other: Non-purified gluten (containing ATIs); Other: Nocebo
- ATIs, nocebo, gluten (Experimental): Participants will start on 1 week of muesli bars with non-purified gluten (containing ATIs) followed by 14 days washout. They will then take 1 week of nocebo muesli bars (containing nothing) followed by 14 days of washout. Finally, they will have 1 week of muesli bars with purified gluten.
  Interventions: Other: Purified gluten; Other: Non-purified gluten (containing ATIs); Other: Nocebo
- Nocebo, ATIs, gluten (Experimental): Participants will start on 1 week of nocebo muesli bars (with nothing) followed by 14 days washout. They will then take 1 week of muesli bars containing non-purified gluten (containing ATIs) followed by 14 days of washout. Finally, they will have 1 week of muesli bars with purified gluten.
  Interventions: Other: Purified gluten; Other: Non-purified gluten (containing ATIs); Other: Nocebo
- Nocebo, gluten, ATIs (Experimental): Participants will start on 1 week of nocebo muesli bars (with nothing) followed by 14 days washout. They will then take 1 week of muesli bars with purified gluten followed by 14 days of washout. Finally, they will have 1 week of muesli bars with non-purified gluten (containing ATIs).
  Interventions: Other: Purified gluten; Other: Non-purified gluten (containing ATIs); Other: Nocebo

INTERVENTIONS:
Other: Purified gluten — 1 low FODMAPs, vegan muesli bar containing purified gluten per day for 1 week, for a total of 10 g purified gluten per day.
Other: Non-purified gluten (containing ATIs) — 1 low FODMAPs, vegan muesli bar containing whole wheat flour with non-purified gluten per day for 1 week, for a total of 10 g non-purified gluten per day.
Other: Nocebo — 1 gluten-free, ATI-free, low FODMAPs, vegan muesli bar per day for 1 week. This is a nocebo because we expect that participants will feel worse even though there is no potential irritant.

SUMMARY:
This crossover randomized controlled trial will evaluate the effects of gluten and gluten combined with amylase-trypsin inhibitors (ATIs) on inducing intestinal and extra-intestinal symptoms in irritable bowel syndrome (IBS) patients. All participants will be put on a gluten-free diet and then challenged with muesli bars containing either purified gluten, gluten with ATIs, or nocebo.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a heterogenous, common gastrointestinal disorder characterized by chronic abdominal pain and altered bowel habits. Many IBS patients report symptom relief on a gluten-free diet (GFD), but it is uncertain whether gluten is the true culprit. The gluten-containing grains wheat, rye, and barley all contain amylase-trypsin inhibitors (ATIs), and a GFD is virtually ATI-free.

This double-blinded crossover randomized controlled trial aims to determine which IBS patients are affected by pure gluten and which are affected by gluten combined with ATIs. IBS patients who respond to and have been on a GFD for 3+ weeks will be randomized to receive a dietary challenge of muesli bars containing either 1) pure gluten, 2) non-purified gluten (containing ATIs), 3) or nocebo for a week followed by a 14 day washout. This will be repeated until all participants have had each dietary challenge.

The study will evaluate the effects and potential mechanisms of purified and non-purified gluten on intestinal and extra-intestinal symptoms in IBS. It is likely that some IBS patients respond to gluten, while others respond to gluten combined with ATIs. Thus, this project may lead to better diagnosis and individualized dietary treatments for IBS.

ELIGIBILITY:
Inclusion Criteria:

* IBS diagnosis based on Rome IV criteria.
* Asymptomatic on a gluten-free diet (IBS-SSS score 0-74).
* Compliance with the study procedures (according to the investigator's own judgement).
* Signing the Study Informed Consent form.

Exclusion Criteria:

* Concurrent systemic disease and/or laboratory abnormalities considered by investigators to be risky or that could interfere with data collection.
* Concurrent organic gastrointestinal disease (i.e. Celiac disease, Inflammatory Bowel Disease, peptic ulcer disease, etc.) other than benign polyps, diverticulosis, hemorrhoids, lipoma and melanosis coli.
* Major abdominal surgery with the exception of hernia repair, appendectomy, Caesarian section, tubal ligation, cholecystectomy, hysterectomy, and hemorrhoidectomy.
* History of active cancer in the last 5 years, other than skin basal cells cancer.
* Pregnant or breastfeeding women.
* Current use of antibiotics or antibiotic treatment within 1 months before the first visit.
* Consumption of probiotics within 1 month prior to the first visit.
* Use of non-authorized medications (see Unauthorized Medications section).
* Patients on a high fibre diet (>35 g/day for males, > 25 g/day for females), consuming high inulin containing foods (>5 g/day), and/or consuming dietary fibre supplements (as assessed by dietary assessment questionnaire) in the 4 weeks prior to the first visit.
* Patients currently participating or having participated in a trial within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome (IBS) symptoms | 1 week gluten or gluten+ATIs intervention compared to nocebo
  Change in IBS symptoms (using Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) during dietary challenge compared to nocebo. The overall score ranges from 0-500 in total, with each of the 5 questions ranging from 0 to 100. A higher score indicates higher symptom severity and the total score is summed.

SECONDARY OUTCOMES:
General gastrointestinal symptoms | 1 week gluten or gluten+ATIs intervention compared to nocebo
  Change in general gastrointestinal symptoms (using The Patient-Reported Outcomes Measurement Information System (PROMIS Scales) for belly pain, diarrhea, constipation, or gas & bloating) during dietary challenge compared to nocebo. Scores are calculated using the Scoring Service by Health Measures and range from 20-80, with medians set at 50 and a standard deviation of 10. Higher scores indicate greater symptom severity. Four PROMIS subscales are being used: Gas & Bloating, Diarrhea, Constipation, and Belly Pain. Each subscale follows the T-scale scoring range of 20-80 and will be measured independently.
Orocecal transit | 1 week gluten or gluten+ATIs intervention compared to nocebo
  Change in colonic transit assessed by SHAPE study (radiopaque markers)
Anti-gliadin antibody (AGA) levels | Serum AGAs will be measured at baseline and after the challenge
  Change in AGA levels after gluten and gluten+ATI challenge will be assessed by ELISA
Gut microbiota profiles | 1 week gluten or gluten+ATIs intervention compared to nocebo
  Change in gut microbiota profiles will be assessed using 16S rRNA Illumina sequencing
Genetic predisposition for celiac disease | Patient HLA DQ2/8 status will be measured at baseline
  Patient HLADQ2/8 status will be assessed at baseline
Depression, anxiety and stress | 1 week gluten or gluten+ATIs intervention compared to nocebo
  Change in depression, anxiety, and stress sub-scales during dietary challenge will be assessed by Depression Anxiety Stress Scale (DASS-21). The DASS-21 has 21 questions. The three subscales (depression, anxiety, and stress) will be reported independently and range from 0 to 42, with higher scores indicating greater symptom severity.
Somatic symptoms | 1 week gluten or gluten+ATIs intervention compared to nocebo
  Change in somatic symptoms like fatigue, sleeping trouble, and pain will be assessed using Patient Health Questionnaire (PHQ-15). Scores range from 0 to 30, with greater scores indicating greater severity.
Stool consistency | 1 week gluten or gluten+ATIs intervention compared to nocebo
  Changes in stool consistency will be assessed by Bristol Stool Scale. Types 1 and 2 indicate harder stools, types 3, 4, and 5 are normal, and types 6 and 7 indicate runnier, more liquid stool.
Gluten levels in stool | Procedure will be explained at baseline
  Presence of gluten in stool samples will be tested for diet compliance using Anti-GIP immunochromatographic strips
Diet assessment | Patients will be asked to take pictures of all meals during each of the 1 week diet challenges
  Dietary tracking will be performed using the MealLogger app
IBS symptom duration | Completed daily for 7 days after each diet challenge
  Evaluates symptom duration at the end of the diet challenge using the IBS-SSS. The overall score ranges from 0-500 in total, with each of the 5 questions ranging from 0 to 100. A higher score indicates higher symptom severity and the total score is summed.
Systemic immune reactivity | 1 week gluten or gluten+ATIs intervention compared to nocebo
  Assessment of pro-inflammatory cytokines levels using peripheral blood mononuclear cell stimulation (PBMC) stimulation in a subset of patients

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Bercik, MD, Principal Investigator — McMaster University; Maria Ines Pinto-Sanchez, MD, Study Director — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boivin M. Socioeconomic impact of irritable bowel syndrome in Canada. Can J Gastroenterol. 2001 Oct;15 Suppl B:8B-11B. doi: 10.1155/2001/401309. PMID 11694908
- [Background] Sanger GJ, Alpers DH. Development of drugs for gastrointestinal motor disorders: translating science to clinical need. Neurogastroenterol Motil. 2008 Mar;20(3):177-84. doi: 10.1111/j.1365-2982.2008.01084.x. PMID 18257767
- [Background] Gibson PR, Shepherd SJ. Evidence-based dietary management of functional gastrointestinal symptoms: The FODMAP approach. J Gastroenterol Hepatol. 2010 Feb;25(2):252-8. doi: 10.1111/j.1440-1746.2009.06149.x. PMID 20136989
- [Background] McKenzie YA, Alder A, Anderson W, Wills A, Goddard L, Gulia P, Jankovich E, Mutch P, Reeves LB, Singer A, Lomer MC; Gastroenterology Specialist Group of the British Dietetic Association. British Dietetic Association evidence-based guidelines for the dietary management of irritable bowel syndrome in adults. J Hum Nutr Diet. 2012 Jun;25(3):260-74. doi: 10.1111/j.1365-277X.2012.01242.x. Epub 2012 Apr 10. PMID 22489905
- [Background] Gaesser GA, Angadi SS. Gluten-free diet: imprudent dietary advice for the general population? J Acad Nutr Diet. 2012 Sep;112(9):1330-1333. doi: 10.1016/j.jand.2012.06.009. No abstract available. PMID 22939437
- [Background] El-Chammas K, Danner E. Gluten-free diet in nonceliac disease. Nutr Clin Pract. 2011 Jun;26(3):294-9. doi: 10.1177/0884533611405538. PMID 21586414
- [Background] van Overbeek FM, Uil-Dieterman IG, Mol IW, Kohler-Brands L, Heymans HS, Mulder CJ. The daily gluten intake in relatives of patients with coeliac disease compared with that of the general Dutch population. Eur J Gastroenterol Hepatol. 1997 Nov;9(11):1097-9. doi: 10.1097/00042737-199711000-00013. PMID 9431901
- [Background] Catassi C, Fabiani E, Iacono G, D'Agate C, Francavilla R, Biagi F, Volta U, Accomando S, Picarelli A, De Vitis I, Pianelli G, Gesuita R, Carle F, Mandolesi A, Bearzi I, Fasano A. A prospective, double-blind, placebo-controlled trial to establish a safe gluten threshold for patients with celiac disease. Am J Clin Nutr. 2007 Jan;85(1):160-6. doi: 10.1093/ajcn/85.1.160. PMID 17209192
- [Background] Lebwohl B, Granath F, Ekbom A, Montgomery SM, Murray JA, Rubio-Tapia A, Green PH, Ludvigsson JF. Mucosal healing and mortality in coeliac disease. Aliment Pharmacol Ther. 2013 Feb;37(3):332-9. doi: 10.1111/apt.12164. Epub 2012 Nov 28. PMID 23190299
- [Background] Leonard MM, Sapone A, Catassi C, Fasano A. Celiac Disease and Nonceliac Gluten Sensitivity: A Review. JAMA. 2017 Aug 15;318(7):647-656. doi: 10.1001/jama.2017.9730. PMID 28810029
- [Background] Maiuri L, Picarelli A, Boirivant M, Coletta S, Mazzilli MC, De Vincenzi M, Londei M, Auricchio S. Definition of the initial immunologic modifications upon in vitro gliadin challenge in the small intestine of celiac patients. Gastroenterology. 1996 May;110(5):1368-78. doi: 10.1053/gast.1996.v110.pm8613040.
- [Background] Lammers KM, Lu R, Brownley J, Lu B, Gerard C, Thomas K, Rallabhandi P, Shea-Donohue T, Tamiz A, Alkan S, Netzel-Arnett S, Antalis T, Vogel SN, Fasano A. Gliadin induces an increase in intestinal permeability and zonulin release by binding to the chemokine receptor CXCR3. Gastroenterology. 2008 Jul;135(1):194-204.e3. doi: 10.1053/j.gastro.2008.03.023. Epub 2008 Mar 21. PMID 18485912
- [Background] Caio G, Volta U, Tovoli F, De Giorgio R. Effect of gluten free diet on immune response to gliadin in patients with non-celiac gluten sensitivity. BMC Gastroenterol. 2014 Feb 13;14:26. doi: 10.1186/1471-230X-14-26. PMID 24524388
- [Background] Ferch CC, Chey WD. Irritable bowel syndrome and gluten sensitivity without celiac disease: separating the wheat from the chaff. Gastroenterology. 2012 Mar;142(3):664-6. doi: 10.1053/j.gastro.2012.01.020. Epub 2012 Jan 24. No abstract available. PMID 22281277
- [Background] Verdu EF. Editorial: Can gluten contribute to irritable bowel syndrome? Am J Gastroenterol. 2011 Mar;106(3):516-8. doi: 10.1038/ajg.2010.490. PMID 21378766
- [Background] Eswaran S, Tack J, Chey WD. Food: the forgotten factor in the irritable bowel syndrome. Gastroenterol Clin North Am. 2011 Mar;40(1):141-62. doi: 10.1016/j.gtc.2010.12.012. PMID 21333905
- [Background] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Background] Verdu EF, Huang X, Natividad J, Lu J, Blennerhassett PA, David CS, McKay DM, Murray JA. Gliadin-dependent neuromuscular and epithelial secretory responses in gluten-sensitive HLA-DQ8 transgenic mice. Am J Physiol Gastrointest Liver Physiol. 2008 Jan;294(1):G217-25. doi: 10.1152/ajpgi.00225.2007. Epub 2007 Nov 15. PMID 18006603
- [Background] Biesiekierski JR, Newnham ED, Irving PM, Barrett JS, Haines M, Doecke JD, Shepherd SJ, Muir JG, Gibson PR. Gluten causes gastrointestinal symptoms in subjects without celiac disease: a double-blind randomized placebo-controlled trial. Am J Gastroenterol. 2011 Mar;106(3):508-14; quiz 515. doi: 10.1038/ajg.2010.487. Epub 2011 Jan 11. PMID 21224837
- [Background] Wahnschaffe U, Schulzke JD, Zeitz M, Ullrich R. Predictors of clinical response to gluten-free diet in patients diagnosed with diarrhea-predominant irritable bowel syndrome. Clin Gastroenterol Hepatol. 2007 Jul;5(7):844-50; quiz 769. doi: 10.1016/j.cgh.2007.03.021. Epub 2007 Jun 5. PMID 17553753
- [Background] Schuppan D, Pickert G, Ashfaq-Khan M, Zevallos V. Non-celiac wheat sensitivity: differential diagnosis, triggers and implications. Best Pract Res Clin Gastroenterol. 2015 Jun;29(3):469-76. doi: 10.1016/j.bpg.2015.04.002. Epub 2015 May 8. PMID 26060111
- [Background] Zevallos VF, Raker V, Tenzer S, Jimenez-Calvente C, Ashfaq-Khan M, Russel N, Pickert G, Schild H, Steinbrink K, Schuppan D. Nutritional Wheat Amylase-Trypsin Inhibitors Promote Intestinal Inflammation via Activation of Myeloid Cells. Gastroenterology. 2017 Apr;152(5):1100-1113.e12. doi: 10.1053/j.gastro.2016.12.006. Epub 2016 Dec 16. PMID 27993525
- [Background] Major G, Pritchard S, Murray K, Alappadan JP, Hoad CL, Marciani L, Gowland P, Spiller R. Colon Hypersensitivity to Distension, Rather Than Excessive Gas Production, Produces Carbohydrate-Related Symptoms in Individuals With Irritable Bowel Syndrome. Gastroenterology. 2017 Jan;152(1):124-133.e2. doi: 10.1053/j.gastro.2016.09.062. Epub 2016 Oct 14. PMID 27746233
- [Background] Wilson B, Whelan K. Prebiotic inulin-type fructans and galacto-oligosaccharides: definition, specificity, function, and application in gastrointestinal disorders. J Gastroenterol Hepatol. 2017 Mar;32 Suppl 1:64-68. doi: 10.1111/jgh.13700. PMID 28244671
- [Background] Spiller R. How do FODMAPs work? J Gastroenterol Hepatol. 2017 Mar;32 Suppl 1:36-39. doi: 10.1111/jgh.13694. PMID 28244663
- [Background] Junker Y, Zeissig S, Kim SJ, Barisani D, Wieser H, Leffler DA, Zevallos V, Libermann TA, Dillon S, Freitag TL, Kelly CP, Schuppan D. Wheat amylase trypsin inhibitors drive intestinal inflammation via activation of toll-like receptor 4. J Exp Med. 2012 Dec 17;209(13):2395-408. doi: 10.1084/jem.20102660. Epub 2012 Dec 3. PMID 23209313
- [Background] El-Salhy M, Ostgaard H, Gundersen D, Hatlebakk JG, Hausken T. The role of diet in the pathogenesis and management of irritable bowel syndrome (Review). Int J Mol Med. 2012 May;29(5):723-31. doi: 10.3892/ijmm.2012.926. Epub 2012 Feb 24. PMID 22366773
- [Background] Mitchell CM, Drossman DA. Survey of the AGA membership relating to patients with functional gastrointestinal disorders. Gastroenterology. 1987 May;92(5 Pt 1):1282-4. doi: 10.1016/s0016-5085(87)91099-7. No abstract available. PMID 3557021
- [Background] Pietzak M. Celiac disease, wheat allergy, and gluten sensitivity: when gluten free is not a fad. JPEN J Parenter Enteral Nutr. 2012 Jan;36(1 Suppl):68S-75S. doi: 10.1177/0148607111426276. PMID 22237879
- [Background] Marcason W. Is there evidence to support the claim that a gluten-free diet should be used for weight loss? J Am Diet Assoc. 2011 Nov;111(11):1786. doi: 10.1016/j.jada.2011.09.030. No abstract available. PMID 22027062
- [Background] Higgins JA. Whole grains, legumes, and the subsequent meal effect: implications for blood glucose control and the role of fermentation. J Nutr Metab. 2012;2012:829238. doi: 10.1155/2012/829238. Epub 2011 Oct 30. PMID 22132324
- [Background] Rosen LA, Ostman EM, Shewry PR, Ward JL, Andersson AA, Piironen V, Lampi AM, Rakszegi M, Bedo Z, Bjorck IM. Postprandial glycemia, insulinemia, and satiety responses in healthy subjects after whole grain rye bread made from different rye varieties. 1. J Agric Food Chem. 2011 Nov 23;59(22):12139-48. doi: 10.1021/jf2019825. Epub 2011 Oct 31. PMID 21961929
- [Background] Russo F, Riezzo G, Chiloiro M, De Michele G, Chimienti G, Marconi E, D'Attoma B, Linsalata M, Clemente C. Metabolic effects of a diet with inulin-enriched pasta in healthy young volunteers. Curr Pharm Des. 2010;16(7):825-31. doi: 10.2174/138161210790883570. PMID 20388093
- [Background] Harris KA, Kris-Etherton PM. Effects of whole grains on coronary heart disease risk. Curr Atheroscler Rep. 2010 Nov;12(6):368-76. doi: 10.1007/s11883-010-0136-1. PMID 20820954
- [Background] Kelly G. Inulin-type prebiotics: a review. (Part 2). Altern Med Rev. 2009 Mar;14(1):36-55. PMID 19364192
- [Background] Abrams SA, Griffin IJ, Hawthorne KM, Liang L, Gunn SK, Darlington G, Ellis KJ. A combination of prebiotic short- and long-chain inulin-type fructans enhances calcium absorption and bone mineralization in young adolescents. Am J Clin Nutr. 2005 Aug;82(2):471-6. doi: 10.1093/ajcn.82.2.471. PMID 16087995
- [Background] Reddy BR. Noncaloric Benefits of Carbohydrates. Nestle Nutr Inst Workshop Ser. 2015;82:27-37. doi: 10.1159/000381999. Epub 2015 Oct 20. PMID 26545117
- [Background] Tarini J, Wolever TM. The fermentable fibre inulin increases postprandial serum short-chain fatty acids and reduces free-fatty acids and ghrelin in healthy subjects. Appl Physiol Nutr Metab. 2010 Feb;35(1):9-16. doi: 10.1139/H09-119. PMID 20130660
- [Background] Neyrinck AM, Delzenne NM. Potential interest of gut microbial changes induced by non-digestible carbohydrates of wheat in the management of obesity and related disorders. Curr Opin Clin Nutr Metab Care. 2010 Nov;13(6):722-8. doi: 10.1097/MCO.0b013e32833ec3fb. PMID 20823777
- [Background] Lee A, Newman JM. Celiac diet: its impact on quality of life. J Am Diet Assoc. 2003 Nov;103(11):1533-5. doi: 10.1016/j.jada.2003.08.027. PMID 14576723
- [Background] Lee AR, Ng DL, Zivin J, Green PH. Economic burden of a gluten-free diet. J Hum Nutr Diet. 2007 Oct;20(5):423-30. doi: 10.1111/j.1365-277X.2007.00763.x. PMID 17845376
- [Background] Verdu EF, Armstrong D, Murray JA. Between celiac disease and irritable bowel syndrome: the "no man's land" of gluten sensitivity. Am J Gastroenterol. 2009 Jun;104(6):1587-94. doi: 10.1038/ajg.2009.188. PMID 19455131
- [Background] Mills EJ, Chan AW, Wu P, Vail A, Guyatt GH, Altman DG. Design, analysis, and presentation of crossover trials. Trials. 2009 Apr 30;10:27. doi: 10.1186/1745-6215-10-27. PMID 19405975
- [Background] Hodge A, Patterson AJ, Brown WJ, Ireland P, Giles G. The Anti Cancer Council of Victoria FFQ: relative validity of nutrient intakes compared with weighed food records in young to middle-aged women in a study of iron supplementation. Aust N Z J Public Health. 2000 Dec;24(6):576-83. doi: 10.1111/j.1467-842x.2000.tb00520.x. PMID 11215004
- [Background] Leffler DA, Dennis M, Edwards George JB, Jamma S, Magge S, Cook EF, Schuppan D, Kelly CP. A simple validated gluten-free diet adherence survey for adults with celiac disease. Clin Gastroenterol Hepatol. 2009 May;7(5):530-6, 536.e1-2. doi: 10.1016/j.cgh.2008.12.032. Epub 2009 Jan 11. PMID 19268725
- [Background] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181
- [Background] Patrick DL, Drossman DA, Frederick IO, DiCesare J, Puder KL. Quality of life in persons with irritable bowel syndrome: development and validation of a new measure. Dig Dis Sci. 1998 Feb;43(2):400-11. doi: 10.1023/a:1018831127942. PMID 9512138
- [Background] Kim ER, Rhee PL. How to interpret a functional or motility test - colon transit study. J Neurogastroenterol Motil. 2012 Jan;18(1):94-9. doi: 10.5056/jnm.2012.18.1.94. Epub 2012 Jan 16. PMID 22323993
- [Background] Megiorni F, Mora B, Bonamico M, Nenna R, Di Pierro M, Catassi C, Drago S, Mazzilli MC. A rapid and sensitive method to detect specific human lymphocyte antigen (HLA) class II alleles associated with celiac disease. Clin Chem Lab Med. 2008;46(2):193-6. doi: 10.1515/CCLM.2008.049. PMID 18076355
- [Background] Zar S, Benson MJ, Kumar D. Food-specific serum IgG4 and IgE titers to common food antigens in irritable bowel syndrome. Am J Gastroenterol. 2005 Jul;100(7):1550-7. doi: 10.1111/j.1572-0241.2005.41348.x. PMID 15984980
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Roalfe AK, Roberts LM, Wilson S. Evaluation of the Birmingham IBS symptom questionnaire. BMC Gastroenterol. 2008 Jul 23;8:30. doi: 10.1186/1471-230X-8-30. PMID 18651941
- [Background] Adam B, Liebregts T, Holtmann G. [Irritable bowel syndrome]. Dtsch Med Wochenschr. 2005 Feb 25;130(8):399-401. doi: 10.1055/s-2005-863064. German. PMID 15717250
- [Background] Fennerty MB. Traditional therapies for irritable bowel syndrome: an evidence-based appraisal. Rev Gastroenterol Disord. 2003;3 Suppl 2:S18-24. PMID 12775999
- [Background] Johanson JF. Options for patients with irritable bowel syndrome: contrasting traditional and novel serotonergic therapies. Neurogastroenterol Motil. 2004 Dec;16(6):701-11. doi: 10.1111/j.1365-2982.2004.00550.x. PMID 15601419
- [Background] Drossman DA, Patrick DL, Whitehead WE, Toner BB, Diamant NE, Hu Y, Jia H, Bangdiwala SI. Further validation of the IBS-QOL: a disease-specific quality-of-life questionnaire. Am J Gastroenterol. 2000 Apr;95(4):999-1007. doi: 10.1111/j.1572-0241.2000.01941.x. PMID 10763950
- [Background] Missbach B, Schwingshackl L, Billmann A, Mystek A, Hickelsberger M, Bauer G, Konig J. Gluten-free food database: the nutritional quality and cost of packaged gluten-free foods. PeerJ. 2015 Oct 22;3:e1337. doi: 10.7717/peerj.1337. eCollection 2015. PMID 26528408
- [Background] Sapone A, Bai JC, Ciacci C, Dolinsek J, Green PH, Hadjivassiliou M, Kaukinen K, Rostami K, Sanders DS, Schumann M, Ullrich R, Villalta D, Volta U, Catassi C, Fasano A. Spectrum of gluten-related disorders: consensus on new nomenclature and classification. BMC Med. 2012 Feb 7;10:13. doi: 10.1186/1741-7015-10-13. PMID 22313950
- [Background] Lionetti E, Catassi C. New clues in celiac disease epidemiology, pathogenesis, clinical manifestations, and treatment. Int Rev Immunol. 2011 Aug;30(4):219-31. doi: 10.3109/08830185.2011.602443. PMID 21787227
- [Background] Natividad JM, Huang X, Slack E, Jury J, Sanz Y, David C, Denou E, Yang P, Murray J, McCoy KD, Verdu EF. Host responses to intestinal microbial antigens in gluten-sensitive mice. PLoS One. 2009 Jul 31;4(7):e6472. doi: 10.1371/journal.pone.0006472. PMID 19649259
- [Background] Bercik P, Denou E, Collins J, Jackson W, Lu J, Jury J, Deng Y, Blennerhassett P, Macri J, McCoy KD, Verdu EF, Collins SM. The intestinal microbiota affect central levels of brain-derived neurotropic factor and behavior in mice. Gastroenterology. 2011 Aug;141(2):599-609, 609.e1-3. doi: 10.1053/j.gastro.2011.04.052. Epub 2011 Apr 30. PMID 21683077
- [Background] Volta U, Pinto-Sanchez MI, Boschetti E, Caio G, De Giorgio R, Verdu EF. Dietary Triggers in Irritable Bowel Syndrome: Is There a Role for Gluten? J Neurogastroenterol Motil. 2016 Oct 30;22(4):547-557. doi: 10.5056/jnm16069. PMID 27426486
- [Derived] Seiler CL, Rueda GH, Miranda PM, Nardelli A, Borojevic R, Hann A, Rahmani S, De Souza R, Caminero A, Curella V, Neerukonda M, Vanner S, Schuppan D, Moayyedi P, Collins SM, Verdu EF, Pinto-Sanchez MI, Bercik P. Effect of gluten and wheat on symptoms and behaviours in adults with irritable bowel syndrome: a single-centre, randomised, double-blind, sham-controlled crossover trial. Lancet Gastroenterol Hepatol. 2025 Sep;10(9):794-805. doi: 10.1016/S2468-1253(25)00090-1. Epub 2025 Jul 21. PMID 40706614